CLINICAL TRIAL: NCT03256942
Title: Evaluation of the Sensitivity of Merz Lips Fullness Assessment Scale Following Etermis 4® Treatment for Lips Volume Augmentation
Acronym: ELISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M900741002
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2017-11

CONDITIONS: Subjects Desiring Lip Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etermis 4® Treatment (Experimental): Etermis 4® will be applied according to the method of administration described in the current version of the Instructions for Use (IFU) until optimal cosmetic result is obtained at the discretion of the treating investigator.
  Single injection session, injections into the lips.
  Interventions: Device: Etermis 4®
- No Treatment (No Intervention)

INTERVENTIONS:
Device: Etermis 4® — Etermis 4® is a sterile non-pyrogenic physiological gel made of reticulated hyaluronic acid (HA) of non-animal origin.
  Arms: Etermis 4® Treatment

SUMMARY:
Primary objective:

- To evaluate the sensitivity of the Merz Lip Fullness Assessment Scale (MLFAS).

Secondary objectives:

* To evaluate the clinical aesthetic improvement outcome in lips appearance four weeks after Etermis 4® injection.
* To evaluate safety/tolerability of Etermis 4® treatment in lips.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female study subjects with thin to medium lips volume (grade 1 to 2 on MLFAS), seeking for hyaluronic acid (HA) for lips volume augmentation in ≥1-point improvement on the MLFAS on both the upper and lower lips and fulfilling the criteria listed in the Instruction for Use (IFU) of the Study Medical Device to be injected.

Exclusion Criteria:

* Subjects with a medical condition and/or medication according to current IFU which is contra indicated for HA filler treatment, or prior facial surgeries or surgical permanent implants, lips augmentation treatment or other aesthetic procedure in the face that could interfere with performance assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Responder rate for treated and for untreated lips at Visit 2 (Week 4), as assessed live by the blinded rater using the Merz Lip Fullness Assessment Scale (MLFAS). | Week 4
  Response is defined as ≥ 1-point improvement on both the upper and lower lips compared to baseline. Upper and lower lips are to be assessed separately.
  The MLFAS is a 5-point scale ranging from 0 (very thin) to 4 (very full). A positive number change from baseline indicates improvement.

SECONDARY OUTCOMES:
Change from baseline for treated and untreated lips at Visit 2 (Week 4) as assessed live by the blinded rater using MLFAS | Week 4
  Upper and lower lips are to be assessed separately. The MLFAS is a 5-point scale ranging from 0 (very thin) to 4 (very full). A positive number change from baseline indicates improvement.
Agreement rate in treated subjects between MLFAS responders and Investigator Global Aesthetic Improvement Scale (Investigator-GAIS) responders at Visit 2 (Week 4). | Week 4
  Agreement for a subject is reached if he/she is a responder for both MLFAS and Investigator-GAIS or he/she is a non-responder for both MLFAS and Investigator-GAIS. GAIS response is defined as at least a "+1 improved" rating on the Investigator -GAIS.
  The MLFAS is a 5-point scale ranging from 0 (very thin) to 4 (very full). A positive number change from baseline indicates improvement. The Investigator-GAIS is a 7-point scale ranging from -3 (very much worse) to +4 (very much improved).
Agreement rate in treated subjects between MLFAS responders and FACE-Q Satisfaction with Lips responders at Visit 2 (week 4). | Week 4
  Agreement for a subject is reached if he/she is a responder for both MLFAS and FACE-Q Satisfaction with Lips or he/she is a non-responder for both MLFAS and FACE-Q Satisfaction with Lips. MLFAS is assessed by a blinded rater. MLFAS response is defined as ≥ 1-point improvement on both the upper and lower lips compared to baseline. FACE-Q Satisfaction with Lips is assessed by the treated subject at baseline and at Visit 2. FACE-Q Satisfaction with Lips response is defined as a positive change in the FACE-Q score.
  The MLFAS is a 5-point scale ranging from 0 (very thin) to 4 (very full). A positive number change from baseline indicates improvement. FACE-Q scores are derived from a questionaire of 10 questions relating to the satisfaction with lips appearance. Answers range from 1 (very dissatisfied) to 4 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (6):
- Germany (6):
  - Dermatologische Privatpraxis, Merz Investigational Site #0490371, Munich, Bavaria
  - Dermatologie München-Neuhausen, Merz Investigational Site #0490372, Munich, Bavaria
  - Haut & Laserzentrum Potsdam, Merz Investigational Site #0490362, Potsdam, Brandenburg
  - Dermatologische Praxis, Merz Investigational Site #0490345, Hamburg, Hanse Stadt Hamburg
  - DRK Kliniken Nordhessen, Merz Investigational Site #0490309, Kassel, Hesse
  - Universität Hamburg, FB Chemie und Molekularbiologie, Merz Investigational Site #0490095, Hamburg

IPD SHARING:
Plan to Share IPD: No